CLINICAL TRIAL: NCT06790277
Title: Effectiveness of Polyurethane Foam (Pink Pad) Compared With Mepilex Dressing for Pressure Ulcer Prevention in Operating Room: A Randomized Control Clinical Trial
Brief Title: Polyurethane Foam-Pink Pad (RCT) Use in OR
Acronym: pink-pad
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah Medical City (Other Government)
Responsible Party: Principal Investigator, Ebtisam Abdellatif Ebrahim Elhihi, Nursing Research and Evidence Based Practice Department, King Abdullah Medical City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-1093; 2323 (Other: SFDA)
Record Dates: First submitted 2024-11-25; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Surgery Subjects; Pressure Ulcer Prevention; Pressure Ulcer of Skin; Pressure Ulcer
Keywords: five layers sacral foam dressing; PINK PAD; pressure ulcers; Patients undergoing cardiac surgery; Mepilex dressing
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyurethane foams (Pink Pad) (Active Comparator): a single use system for use in surgical procedures.it will be used only by operating room nurses Patient will be examined by wound management team after the operation then at day 3- and 7-days post operation.
  Interventions: Device: Polyurethane foams (Pink Pad)
- Mepilex Border Sacrum dressings (Active Comparator): a single use system for use in surgical procedures.it will be used only by operating room nurses Patient will be examined by wound management team after the operation then at day 3- and 7-days post operation.
  Interventions: Device: Mepilex Border Sacrum dressings

INTERVENTIONS:
Device: Mepilex Border Sacrum dressings — Both types of intervention will be available in the operating room. Patient will be examined by head nurse of wound management team after the operation then at day 3- and 7-days post operation. The dressing should be removed after 7 days post operation or if there is any clinical indication for removal. If a patient is discharged before 7 days post operation for any reason the head nurse of wound management team will examine the patient before discharge. Follow up will be for maximum 7 days post operation for each subject. Any patient will be unable to continue the study because of death or change in the care setting will be excluded from the study.
  Arms: Mepilex Border Sacrum dressings
Device: Polyurethane foams (Pink Pad) — Both types of intervention will be available in the operating room. Patient will be examined by head nurse of wound management team after the operation then at day 3- and 7-days post operation. The dressing should be removed after 7 days post operation or if there is any clinical indication for removal. If a patient is discharged before 7 days post operation for any reason the head nurse of wound management team will examine the patient before discharge. Follow up will be for maximum 7 days post operation for each subject. Any patient will be unable to continue the study because of death or change in the care setting will be excluded from the study.
  Arms: Polyurethane foams (Pink Pad)

SUMMARY:
King Abdullah medical city has a cardiac center, and a lot of open-heart surgeries are performed there, and both polyurethane foam (pink Pad) and Mepilex dressing are applied to those patients. Therefore, the present study was designed to compare the effects of polyurethane foam (pink Pad) versus Mepilex dressing for prevention of pressure ulcer in operating room.

DETAILED DESCRIPTION:
There are two types of intervention available in King Abdullah medical city for operating room pressure ulcer prevention. Polyurethane foams (Pink Pad) are a single use system for use in surgical procedures. The system consists of a proprietary formulation for the pink foam pad, non-woven lift sheet, body straps, head rests, and boot liners. It aids hospital facilities in providing a safe and effective method of management of the patient for pressure ulcers and non-movement for patients in the Trendelenburg position.

Mepilex Border Sacrum dressings are self-adherent, multilayer foam dressings designed for use on sacrum aiming to prevent pressure ulcers. The dressings are used in addition to standard care protocols for pressure ulcer prevention.

All included patients received standard PU prevention according to hospital protocols, based on contextualization and adaptation of International guidelines ( European Pressure Ulcer Advisory Panel, 2021 ), which involved: assessment of PU risk through the Braden Scale at hospital admission,

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18.
* Willing to participate.
* Patients undergoing cardiac surgery.
* Patient who is at risk for PU development as measured with Braden scale.
* Patient who has skin intact and having a life expectancy greater than 72 hours as per clinical judgement.

Exclusion Criteria:

* Subjects under 17
* Not consenting to participate
* Patients with suspected hypersensitivity reactions to any of the dressing formulation's ingredients.
* Patients who are unable to continue the study because of death or change in the care setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Pressure ulcer incidence | 7 days
  Pressure ulcer incidence will be assessed by using Bates-Jensen Wound Assessment Tool (BWAT) after operation then day 3 and day 7 for both treatments.

SECONDARY OUTCOMES:
occurrence of pressure ulcer | 7 days
  The occurrence of pressure ulcer will be documented in data collection then calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulla Medical City in Holy capital, Mecca, Western Reagan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) will not be shared , but the data can be reviewed by regulatory officer

REFERENCES:
- [Derived] Elhihi EA, Almuwallad SA, Alqrashi BM, Nada EM, Alduaiji NA, Alfakeeh AA. Effectiveness of a Single-Use Polyurethane Foam Positioning Pad Compared With Five-Layer Foam Sacral Dressing for Pressure Ulcer Prevention in the Operating Room: A Randomized Controlled Clinical Trial. Health Sci Rep. 2025 Aug 10;8(8):e70963. doi: 10.1002/hsr2.70963. eCollection 2025 Aug. PMID 40791282

DOCUMENTS (2):
  • Study Protocol (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT06790277/Prot_000.pdf
  • Informed Consent Form (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT06790277/ICF_001.pdf